CLINICAL TRIAL: NCT01840111
Title: Environments as Smoking Cues: Imaging Brain Substrates, Developing New Treatments
Brief Title: Environments as Smoking Cues: Imaging Brain Substrates, Developing New Treatments (CameraCue)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00033975
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Smoking; Healthy
Keywords: smoking environment; cue-exposure; cigarettes; nicotine; fMRI
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Quit Smoking 6 hours — participants will quit smoking 6 hours prior to the cue-exposure sessions
Behavioral: Quit Smoking 24 hours — participants will quit smoking 24 hours prior to the fMRI scan

SUMMARY:
The overarching goals of this proposal are to 1) identify the network of brain regions specifically activated by personal smoking environment cues and 2) to evaluate the effects of exposure to these cues on smoke self-administration and subjective reactivity. The results of this study will inform the development of novel and more efficacious cue-exposures therapies targeted at helping smokers quit smoking and will provide novel mechanism information regarding the influence of environmental context on drug taking.

The investigator hypothesizes that cue-exposure treatments (CETs), in which drug use is prevented during exposure to drug cues (e.g. lit cigarette) have been of limited efficacy in part because they have not included cues representative of the contexts in which drug use occurs. By demonstrating that context cues have a differential and robust influence on brain and behavioral responses, we will have provided a substantial basis for including such stimuli in the context of treatment. At the same time, we will have identified novel mechanisms by which such stimuli promote continued drug use and relapse.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* between the ages of 18 and 55
* smoking an average of 5 cigarettes per day for at least one year
* breath CO (carbon monoxide) level > 8 ppm (if ≤ 8 ppm, then NicAlert Strip > 2)
* no interest in quitting smoking for the duration of time required for the experiment
* right-handed as measured by a three-item scale used in our laboratory
* ability to identify 4 personal smoking and 4 personal non-smoking places

Exclusion Criteria:

* inability to attend all required experimental sessions
* significant health problems
* use of psychoactive medications
* use of smokeless tobacco
* current alcohol or drug abuse
* use of illegal drugs as measured by urine drug screen
* current use of nicotine replacement therapy or other smoking cessation treatment
* presence of conditions that would make MRI unsafe (e.g., pacemaker)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Signal Change in Functional Magnetic Resonance Imaging (fMRI) BOLD Signal between Personal Environment Pictures Relative to Standard Environment Pictures | following 24 hours of smoking abstinence
  During fMRI scanning participants will view pictures of personal and standard smoking and non-smoking environments; and also pictures of smoking-related and non-smoking related objects

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McClernon, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] McClernon FJ, Conklin CA, Kozink RV, Adcock RA, Sweitzer MM, Addicott MA, Chou YH, Chen NK, Hallyburton MB, DeVito AM. Hippocampal and Insular Response to Smoking-Related Environments: Neuroimaging Evidence for Drug-Context Effects in Nicotine Dependence. Neuropsychopharmacology. 2016 Feb;41(3):877-85. doi: 10.1038/npp.2015.214. Epub 2015 Jul 16. PMID 26179147